CLINICAL TRIAL: NCT05840809
Title: Pharmacokinetics of Drugs Used to Treat Drug-sensitive Tuberculosis in Breastfeeding Mother-infant Pairs: An Observational Pharmacokinetic Study
Brief Title: Pharmacokinetics of Drugs Used to Treat Drug Sensitive Tuberculosis in Breastfeeding Mother-infant Pairs
Acronym: MILK TB
Status: Active, not recruiting | Type: Observational
Sponsor: University of Liverpool (Other)
Collaborators: Makerere University (Other)
Responsible Party: Principal Investigator, Catriona Waitt, Professor Catriona Waitt, University of Liverpool
Other Study IDs: MILK TB
Record Dates: First submitted 2023-04-10; First posted 2023-05-03 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Tuberculosis Active; Breastfeeding; Tuberculosis
Keywords: Breastfeeding; Tuberculosis; Pharmacokinetic
MeSH Terms: conditions — Tuberculosis; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples will be retained until all pharmacokinetic bioanalysis is complete
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Women who require first-line treatment for drug-sensitive tuberculosis whilst breastfeeding and their babies.
  This regimen consists of rifampicin, isoniazid, ethambutol and pyrazinamide for 2 months (intensive phase) followed by a further four months of rifampicin and isoniazid (continuation phase)
  Interventions: Drug: First line tuberculosis treatment

INTERVENTIONS:
Drug: First line tuberculosis treatment — This is an observational study - the decision to use first-line tuberculosis treatment will have already been made by the responsible clinician. The study itself does not require any additional intervention.

SUMMARY:
Pregnant or lactating women requiring treatment for drug sensitive-TB will be identified and invited for sampling. If they are pregnant when identified, they will be invited for sampling after delivery. Plasma and breastmilk samples will be obtained pre-dose and at 2, 4, 6, and 8 hours post-dose. If logistics permit (for example living close to the research unit), the participant will be invited for a further sample at 24 hours post-dose. A heelprick sample will also be obtained from their breastfed infants at maternal trough (prior to maternal dose) and at a random timepoint (once per infant) over the 8-hour pharmacokinetic sampling visit in order to characterize concentrations of these drugs over an 8-hour dosing interval. Total concentrations of plasma and breastmilk Isoniazid, Rifampicin, Pyrazinamide and Ethambutol will be determined.

If a participant has her first pharmacokinetic profile in the intensive phase of TB treatment (whilst on all four of isoniazid, rifampicin, pyrazinamide and ethambutol), she will be invited for a subsequent sampling day with the same time points when she is on the continuation phase of therapy (rifampicin and isoniazid).

DETAILED DESCRIPTION:
Background

Worldwide, ~50% of women take medication during breastfeeding. Data surrounding the exposure of the breastfed infant to drugs and any associated risks are sparse. Despite longstanding recommendations from the US Food and Drug Administration (FDA) for lactation studies to be performed close to licensing for drugs anticipated to be widely used in women of childbearing age, such studies are rarely undertaken. Drugs taken by the breast feeding mother on TB treatment can be passed from the maternal circulation to the milk and then to the breastfed infant, a concern of effects of anti-tuberculosis drugs on nursing infants. Most TB drugs are metabolized by the liver, triggering a potential risk of drug accumulation in infants due to their immature liver function particularly in premature infants.

Drugs are transferred to milk in small quantities, and many have been used without obvious infant toxicity for many years hence the large gaps in the data. Pharmacokinetic (PK) information of anti- TB drugs transfer to breast milk and breastfed infant is crucial to limit the development of drug resistance and understand the safety of prolonged exposure through breast milk.

Problem Statement

Whilst data on TB drug penetration into breastmilk is limited, information on clinically relevant infant exposure to TB drug-sensitive is even more limited and is an important knowledge gap both for safety, and because therapeutic concentrations could be 1) protective in exposed infants, obviating the need for TB preventive therapy or 2) sub- therapeutic concentrations could select for resistance in those infants infected with Mycobacterium tuberculosis.

Recruitment

Women will be identified as they attend the clinic for TB treatment at the IDI and KCCA clinics in Uganda. Should a woman express willingness to participate, once eligibility for enrolment in the study has been determined, informed consent will be obtained.

Pharmacokinetic Study Day

On arrival, an intravenous cannula will be inserted into the antecubital fossa, and samples taken for trough drug measurement. After a standardized breakfast the participant will be administered standard doses of the prescribed medication. Blood samples will be collected at 2, 4, 6, 8 and ideally* 24 hours. Advice to freely breastfeed the baby will be given. The participant will be asked to provide a 2-5 ml sample of expressed breast milk pre-dose, and at 2, 4, 6 and 8 hours post dosing. A blood sample from the infant will be collected at maternal trough (pre-dose) and at a 3-8 hours post maternal dose (the second time point will be allocated sequentially to ensure spread of datapoints). The mother will be administered a standard lunch.

*Due to the logistic considerations of sampling a postpartum mother and her infant who may have travelled a long distance to the clinic, the 24-hour sample may not be collected in all cases.

Maternal albumin and creatinine will be sampled as they are important for isoniazid exposure. Maternal questionnaires will be filled on each visit to assess depression and anxiety; Generalised anxiety disorder questionnaire (GAD-7), Patient health questionnaire (PHQ-9), and the Beliefs about medicines questionnaire (BMQ). Infant clinical assessment will include use of the Gross Motor Development (GMD) checklist

Sample Size Determination

This study is exploratory, as no prior study has characterized the exposure of these drugs in maternal plasma, breastmilk and infant plasma. There are no prior data upon which to build a sample size calculation, and there is no comparison between groups which requires statistical analysis with a pre-specified certainty.

Since no information is available about the penetration of these drugs into breastmilk, the following approach was used, described in detail for rifampicin.

A previously published pop-PK model of rifampicin in plasma was modified, adding a compartment to describe breastmilk concentrations. This was characterised using an approach similar to an effect compartment described by a time delay and an accumulation ratio between breastmilk and plasma. The half-life of the delay was fixed to 1 h and the accumulation ratio to 1.5, with 30% between-subject variability in both parameters. These were chosen to mimic a PK profile similar to Waitt et al. It was assumed that there would be 15 individuals (considering a mother-infant dyad as a single unit) with an intensive PK sampling at 0, 1, 2, 4, 6 and 8 hours post-dose of paired plasma and breastmilk (30% error in the breastmilk measurements was assumed) and Stochastic Simulations and Estimations (SSEs) were performed to evaluate trial design. This design can characterise all the typical values of the plasma PK parameters with precision of better than 11% RSE, and all the breastmilk parameters are well characterised with a precision of 1.14% and 0.591% RSE on delay and accumulation ratio, respectively.

Interim analysis after five participants is part of study design

Analysis of Endpoints

Pharmacokinetic data will be analysed using a population pharmacokinetic approach to estimate pharmacokinetic parameters and produce modelled fits to exposure data. Inter-individual variability will be quantified in relation to the covariates.

Non-compartmental methods will be used to assess correlations between maternal breast milk drug concentrations and measures of drug exposure in the infant (eg AUC) and pharmacodynamic factors.

ELIGIBILITY:
Inclusion Criteria:

1. A personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study.
2. Participants who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Woman is aged 18 years or older
4. Receiving treatment for drug sensitive TB
5. Pregnant or breastfeeding at enrolment

Exclusion Criteria:

1. Severe maternal or infant illness which in the opinion of the patient's clinician would interfere with her participation in the study.
2. Breastfed infant is aged over 12 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breastfeeding women, including those living with HIV, treated for TB will be recruited prospectively from Infectious Diseases clinic (IDI) and IDI Kampala City Council Authority (KCCA) affiliated clinics. The clinics treat pregnant and breast-feeding women infected with TB. We anticipate that 80% of women will be living with HIV. Drug-drug interactions between antiretroviral therapy (ART) and TB drugs could affect the exposure of TB drugs. Data on concomitant medication will be recorded and included as a covariate in the pharmacokinetic analysis. In accordance with national protocol, the infants of mothers diagnosed with TB treatment will receive isoniazid preventive therapy for six months (the duration of the mothers' TB treatment).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2026-01-29 (Estimated)

PRIMARY OUTCOMES:
Concentration of rifampicin in maternal plasma | 0-24 hours after maternal dose
  Pharmacokinetic
Concentration of rifampicin in breastmilk | 0-24 hours after maternal dose
  Pharmacokinetic
Concentration of rifampicin in infant plasma | 0-24 hours after maternal dose
  Pharmacokinetic
Concentration of isoniazid in maternal plasma | 0-24 hours after maternal dose
  Pharmacokinetic
Concentration of isoniazid in breastmilk | 0-24 hours after maternal dose
  Pharmacokinetic
Concentration of isoniazid in infant plasma | 0-24 hours after maternal dose
  Pharmacokinetic
Concentration of ethambutol in maternal plasma | 0-24 hours after maternal dose
  Pharmacokinetic
Concentration of ethambutol in breastmilk | 0-24 hours after maternal dose
  Pharmacokinetic
Concentration of ethambutol in infant plasma | 0-24 hours after maternal dose
  Pharmacokinetic
Concentration of pyrazinamide in maternal plasma | 0-24 hours after maternal dose
  Pharmacokinetic
Concentration of pyrazinamide in breastmilk | 0-24 hours after maternal dose
  Pharmacokinetic
Concentration of pyrazinamide in infant plasma | 0-24 hours after maternal dose
  Pharmacokinetic

SECONDARY OUTCOMES:
Maximum concentration of rifampicin in maternal plasma | 0-24 hours after maternal dose
  Pharmacokinetic measurement
Maximum concentration of rifampicin in breastmilk | 0-24 hours after maternal dose
  Pharmacokinetic measurement
Maximum concentration of isoniazid in maternal plasma | 0-24 hours after maternal dose
  Pharmacokinetic measurement
Maximum concentration of isoniazid in breastmilk | 0-24 hours after maternal dose
  Pharmacokinetic measurement
Maximum concentration of ethambutol in maternal plasma | 0-24 hours after maternal dose
  Pharmacokinetic measurement
Maximum concentration of ethambutol in breastmilk | 0-24 hours after maternal dose
  Pharmacokinetic measurement
Maximum concentration of pyrazinamide in maternal plasma | 0-24 hours after maternal dose
  Pharmacokinetic measurement
Maximum concentration of pyrazinamide in breastmilk | 0-24 hours after maternal dose
  Pharmacokinetic measurement
Anxiety in mothers | During pharmacokinetic study visits (up to 52 weeks postpartum)
  Generalised anxiety disorder (GAD7 questionnaire)
Depression in mothers | During pharmacokinetic study visits (up to 52 weeks postpartum)
  Patient health questionnaire (PHQ-9)
Maternal beliefs about medicines | During pharmacokinetic study visits (up to 52 weeks postpartum)
  Beliefs about Medicines Questionnaire (BMQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Infectious Diseases Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data (drug concentrations) will be made available through an online repository such as Zeonodo
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Protocol, SAP and ICF will shortly become available. Anonymised datasets will become available after primary analysis
Access Criteria: Permissions to access the documents and datasets can be requested via the MILK Zenodo Community.
URL: https://zenodo.org/record/7798349#.ZDQH_HtByUk

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT05840809/Prot_SAP_000.pdf